CLINICAL TRIAL: NCT04178681
Title: The Effects of Different Fat Structures on Postprandial Responses in Healthy Subjects
Brief Title: Postprandial Effects of Milk Fats
Acronym: POEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wageningen University (Other)
Collaborators: Friesland Campina (Unknown)
Responsible Party: Principal Investigator, Lydia A. Afman, Principal Investigator, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL69492.081.19
Record Dates: First submitted 2019-08-16; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Genomics; Postprandial Metabolism; Nutrition; Metabolism
Keywords: Humans; Milk fat; Clinical Trial; Genomics; Metabolism; Nutrition

STUDY DESIGN:
Intervention Model Description: Each research subject will visit the university on three separate occasions with a wash-out period of at least one week. At each visit the research subject will undergo one of the three dietary lipid challenge tests (a shake) in a randomized order. All research subjects have consumed all three dietary lipid challenge tests at the end of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- V-A-C (Experimental): Order of administration:
  1. 100% vegetable fat blend
  2. 100% Anhydrous Milk Fat (AMF)
  3. 100% Cream (AMF + milk fat globular membranes)
  Interventions: Other: 100% vegetable blend; Other: 100% AMF; Other: 100% cream
- V-C-A (Experimental): Order of administration:
  1. 100% vegetable fat blend
  2. 100% Cream (AMF + milk fat globular membranes)
  3. 100% Anhydrous Milk Fat (AMF)
  Interventions: Other: 100% vegetable blend; Other: 100% AMF; Other: 100% cream
- A-V-C (Experimental): Order of administration:
  1. 100% Anhydrous Milk Fat (AMF)
  2. 100% vegetable fat blend
  3. 100% Cream (AMF + milk fat globular membranes)
  Interventions: Other: 100% vegetable blend; Other: 100% AMF; Other: 100% cream
- A-C-V (Experimental): Order of administration:
  1. 100% Anhydrous Milk Fat (AMF)
  2. 100% Cream (AMF + milk fat globular membranes)
  3. 100% vegetable fat blend
  Interventions: Other: 100% vegetable blend; Other: 100% AMF; Other: 100% cream
- C-A-V (Experimental): Order of administration:
  1. 100% Cream (AMF + milk fat globular membranes)
  2. 100% Anhydrous Milk Fat (AMF)
  3. 100% vegetable fat blend
  Interventions: Other: 100% vegetable blend; Other: 100% AMF; Other: 100% cream
- C-V-A (Experimental): Order of administration:
  1. 100% Cream (AMF + milk fat globular membranes)
  2. 100% vegetable fat blend
  3. 100% Anhydrous Milk Fat (AMF)
  Interventions: Other: 100% vegetable blend; Other: 100% AMF; Other: 100% cream

INTERVENTIONS:
Other: 100% vegetable blend — Dietary lipid challenge test: 600 ml skimmed milk plus 95 gram of vegetable fat blend.
Other: 100% AMF — Dietary lipid challenge test: 600 ml skimmed milk plus 95 gram of anhydrous milk fat.
Other: 100% cream — Dietary lipid challenge test: 600 ml skimmed milk plus 95 gram of anhydrous milk fat plus milk fat globular membranes.

SUMMARY:
Nowadays, mostly vegetable fat blends are used in infant formula, but the use of bovine milk fat is increasing. In terms of fat structure, bovine milk fat and vegetable fats differ. Bovine milk fat has a higher percentage of palmitic acid attached to the sn-2 position of the glycerol backbone compared to vegetable fat blend. Also bovine milk fat contains milk fat globular membranes, as opposed to vegetable fat. With this study the investigators want to examine the effects of a vegetable fat blend versus bovine milk fat without globular membranes and bovine milk fat with globular membranes on underlying mechanistic, immune and metabolic responses.

DETAILED DESCRIPTION:
Rationale: Human milk is considered as the ideal food for full-term infants. The composition and function of human milk is unique and has provided the basis for the development of modern artificial milk formulas that mimic its complex biological positive effects on infants and can provide an appropriate substitute for non-breastfed infants. An important component in human milk are the lipids, as they deliver 50% of the total energy to infants. Nowadays, mostly vegetable fat blends are used in infant formula, but the use of bovine milk fat is increasing. In terms of fat structure, bovine milk fat and vegetable fats differ. Bovine milk fat has a higher percentage of palmitic acid attached to the sn-2 position of the glycerol backbone compared to vegetable fat blend. Also bovine milk fat contains milk fat globular membranes, as opposed to vegetable fat. Knowledge on how these differences influence underlying mechanistic, immune and metabolic responses is lacking.

Objectives: The primary objective of this study is to determine the effect of three different fat blends on underlying mechanistic and immune responses in the circulation. The secondary objectives of this study are: 1) to examine the effects of the three different fat blends on postprandial triglyceride concentration and other cardio-metabolic markers in the circulation, 2) to investigate the effect of the three different fat blends on postprandial feelings of hunger and satiety, and 3) to investigate how comparable cytokine measurements are in blood samples obtained via a catheter cannula compared to cytokine measurements in dried blood spots obtained via a finger prick.

Study design: The POEMI Study is a double-blind randomized cross-over acute intervention study in which each research subject will visit the university on three separate occasions with a wash-out period of at least one week. At each visit the research subject will undergo one of the three dietary lipid challenge tests (a shake) in a randomized order. On each study day research subjects will be asked to clock in 30 minutes prior to the first data collection points and a catheter cannula will be inserted in a antecubital vein. After the 30 minute rest, blood will be drawn from the catheter cannula and via a finger prick (baseline measurements, t0). After the baseline measurements, the research subjects will have to consume the shake within a time frame of 10 minutes. Blood is again drawn from the catheter cannula at t= 1, 2, 3, 4, 5, 6, 7, and 8 hours after consumption, with an additional finger prick at t=6. A questionnaire on hunger and satiety feelings will be taken after every blood draw.

Study population: The base population will consist of 40 healthy men and women with a BMI ranging from 22 to 27 kg/m2, aged 40 to 70 years old, selected from the surroundings of Wageningen through the mailing list for potential study research subjects of the division of Human Nutrition and health of Wageningen University. If needed, additional recruitment of research subjects will take place by flyers and posters, or advertisements in local newspapers.

Intervention: The dietary lipid challenge tests will be provided in the form of a liquid shake (0.6 L). Each shake will contain 95 gram of fat. The three types of fat that will be tested include: a) 100% vegetable fat blend, b) 100% Anhydrous milk fat (AMF), c) 100% cream (AMF + milk fat globular membranes).

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy man or woman
* Age 40-70y at the time of recruitment
* BMI of 22-27 kg/m2
* Having a Hb value above 8.4 (men) or 7.4 (women) mmol/L (will be checked at the screening visit)
* Having veins suitable for blood sampling via a catheter cannula (judged by study nurse/ medical doctor)
* Having a general practitioner
* Signed informed consent

Exclusion Criteria:

* Any chronic metabolic, gastrointestinal, inflammatory or chronic disease (such as diabetes, anaemia, hepatitis, cardiovascular disease)
* History of gastro-intestinal surgery or having (serious) gastro-intestinal complaints
* Renal or hepatic malfunctioning (pre-diagnosis or determined based on ALAT, ASAT and creatinine values)
* Use of medication that may influence the study results, such as laxatives, stomach protectors and drugs that can affect intestinal motility.
* Donated or intend to donate blood from 2 months before the study until the end of the study
* Reported slimming, medically prescribed or vegan diet
* Unstable body weight (weight gain or loss >5 kg in the past three months)
* Current smokers
* Alcohol on average: more than 2 consumptions/day or more than 14 consumptions/week
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported)
* Use of illicit drugs
* Food allergies for products that the investigators use in the study
* Participation in another clinical trial at the same time, or in the month preceding the start of this study
* Inability to understand study information and/or communicate with staff
* Members of the research team
* Working, or doing an internship or thesis at the division "Human Nutrition and Health", Wageningen University

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-02 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in transcriptomics from baseline to 6 hours after consumption of the three different fat blends, to elucidate underlying mechanistic responses in the circulation. | Baseline and 6 hours after consumption of the dietary lipid challenge.
  By using untargeted whole genome Affymetrix microarray the investigators will measure gene expression in isolated monocytes.
Change in cytokine concentration from baseline and every hour until 8 hours after consumption of the different fat blends, to elucidate the effect on immune responses in the circulation. | Baseline and every hour until 8 hours after consumption of the dietary lipid challenge.
  Cytokine concentrations in the circulation will be measured via ELISA.
Change in functional responses to LPS stimulation of isolated monocytes from the circulation from baseline to 6 hours after consumption of the different fat blends. | Baseline and 6 hours after consumption of the dietary lipid challenge.
  Cell study with isolated monocytes from the circulation. The cells will be treated with LPS to evaluate functional responses. We will measure fold changes.
Change in sensitivity of isolated monocytes from the circulation. | Baseline and 6 hours after consumption of the dietary lipid challenge.
  Cell study with isolated monocytes from the circulation. The cells will be treated with different fat loads and inflammatory stimuli to evaluate the sensitivity of the collected monocytes. We will measure fold changes.

SECONDARY OUTCOMES:
Postprandial triacylglycerol changes | Baseline and every hour until 8 hours after consumption of the dietary lipid challenge.
  TAG concentration in plasma will be measured in a clinical chemical lab.
Postprandial glucose changes | Baseline and every hour until 8 hours after consumption of the dietary lipid challenge.
  Cardio-metabolic markers such as glucose (mg/dl) will be measured in the circulation.
Postprandial adiponectin changes | Baseline and every hour until 8 hours after consumption of the dietary lipid challenge.
  Cardio-metabolic markers such as adiponectin (pg/ml) will be measured in the circulation.
Postprandial insulin changes | Baseline and every hour until 8 hours after consumption of the dietary lipid challenge.
  Cardio-metabolic markers such as insulin (mIU/L) will be measured in the circulation.
Postprandial (untargeted) protein profile changes | Baseline and every hour until 8 hours after consumption of the dietary lipid challenge.
  Using untargeted proteomic platforms, the changes in protein profiles in the circulation will be measured.
Postprandial (targeted) protein profile changes | Baseline and every hour until 8 hours after consumption of the dietary lipid challenge.
  Using targeted proteomic platforms, the changes in protein profiles in the circulation will be measured.
Postprandial (untargeted) metabolite profile changes | Baseline and every hour until 8 hours after consumption of the dietary lipid challenge.
  Using untargeted metabolomic platforms, the changes in protein profiles in the circulation will be measured.
Postprandial (targeted) metabolite profile changes | Baseline and every hour until 8 hours after consumption of the dietary lipid challenge.
  Using targeted metabolomic platforms, the changes in protein profiles in the circulation will be measured.
Postprandial changes in feelings of hunger and satiety | Baseline and every hour until 8 hours after consumption of the dietary lipid challenge.
  Feelings of hunger and satiety will be measured via a questionnaire using a Visual Analog Scale (VAS), a 100 mm line anchored at each end by descriptors. Research subjects will place a mark on the scale that corresponds to their feelings of hunger and satiety. The distance from the lower end of the scale is then measured and recorded.
Cytokine concentration comparison | Baseline and 6 hours after consumption of the dietary lipid challenge.
  Cytokine concentrations in the circulation obtained via catheter cannula will be measured via ELISA. The investigators will also measure cytokine concentrations in dried blood spots obtained via a finger prick (via a Meso Scale Discovery Electrochemiluminescence platform).

OTHER OUTCOMES:
Immune cell populations | Baseline and 6 hours after consumption of the dietary lipid challenge.
  Relative immune cell populations will be determined in whole blood via FACS analysis.
CRP | Before the start of a study day.
  The CRP value of each research subject will be determined by using a QuikRead CRP test.
WHR | Baseline
  Both waist and Hip circumference will be measured using a measuring tape.
BMI | Baseline
  weight (in kg) and height (in meters) will be measured and combined to report BMI in kg/m^2
Habitual intake | Baseline
  As assessed by a validated FFQ.
Renal or hepatic malfunctioning | Baseline
  ALAT (IU/L), ASAT (IU/L) will be measured in a clinical chemical lab.
Renal malfunctioning | Baseline
  creatinine (mg/dL) will be measured in a clinical chemical lab.
Anemia | Baseline
  Hemoglobin will be determined via a finger prick.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Afman, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Collected data will be coded.